CLINICAL TRIAL: NCT00323167
Title: Rare Genetic Disorders of the Airways: Cross-sectional Comparison of Clinical Features, and Development of Novel Screening and Genetic Tests
Brief Title: Rare Genetic Disorders of the Breathing Airways
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Research Resources (NCRR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 05-2979; U54RR019480 (NIH); RDCRN 5902 (Other: UNC)
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Kartagener Syndrome; Cystic Fibrosis; Pseudohypoaldosteronism; Primary Ciliary Dyskinesia
Keywords: Variant Cystic Fibrosis; Primary Ciliary Dyskinesia
MeSH Terms: conditions — Kartagener Syndrome; Cystic Fibrosis; Pseudohypoaldosteronism; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Respiratory cultures, nasal samples, and blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Mucociliary clearance, in which mucus secretions are cleared from the breathing airways, is the primary defense mechanism for the lungs. Inhaled particles, including microbes that can cause infections, are normally entrapped in mucus on the airway surfaces and then cleared out by the coordinated action of tiny hair-like structures called cilia. Individuals with primary ciliary dyskinesia, variant cystic fibrosis, and pseudohypoaldosteronism have defective mucociliary clearance. The purpose of this study is to collect clinical and genetic information about these three airway diseases to improve current diagnostic procedures.

DETAILED DESCRIPTION:
Two types of genetic diseases are associated with abnormal mucociliary clearance. The first type results in defective ciliary function and includes primary ciliary dyskinesia (PCD), also known as Kartagener Syndrome. The second type results in defective ion transportation and includes variant cystic fibrosis (CF) and pseudohypoaldosteronism (PHA). The clinical manifestations of these three diseases overlap, and current evaluation procedures are inadequate for an accurate and timely diagnosis. A delayed diagnosis, coupled with poorly defined disease categories, results in sub-optimal treatment regimens. The purpose of this study is to better define the clinical and genetic features of PCD, variant CF, and PHA to develop improved diagnostic procedures. The study will also compare prevalence and age-related information among the three diseases and classic CF. Outcomes of this study may lead to improved clinical care and novel therapeutic approaches for rare genetic disorders of the airways.

Prior to study entry, previous clinical data on all participants will be reviewed to ensure that individuals do not have common variants of asthma. In some cases, further clinical evaluation (sweat chloride testing, immunodeficiency testing, and a high-resolution computed tomography scan) may be recommended. Eligible participants will attend an initial six-hour study visit similar to a standard diagnostic evaluation. The participant's medical history will be reviewed and a physical examination will include height, weight, and vital sign measurements. Respiratory cultures, nasal samples, and blood will be collected. Non-invasive techniques will be used to measure oxyhemoglobin saturation levels and airflow; a chest x-ray will be required if none has been done in the last six months.

If a firm diagnosis of PCD or variant CF has not been established after completion of the first study visit, the participant may return for additional visits. Salivary and semen samples may be collected from some individuals. A sweat chloride test and nasal potential difference test may also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Received a standard diagnostic evaluation prior to study entry that resulted in one of the following three profiles:

  1. High likelihood of PCD diagnosis, based on ciliary ultrastructural changes seen on electron microscopy or clinical features (chronic sinopulmonary disease, chronic otitis media, history of neonatal respiratory distress or situs inversus) OR one clinical feature of PCD and a sibling with PCD
  2. Chronic sino-pulmonary disease with clinical features that overlap with variant CF and PCD, but with diagnostic tests that rule out classical CF (sweat chloride testing and CF gene mutation screening)
  3. Known or suspected PHA (or variant PHA), possibly including elevated (or borderline) sweat chloride values

Exclusion Criteria:

* Has not received a standard clinical evaluation to rule out other disorders associated with chronic sino-pulmonary disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with suspected primary ciliary dyskinesia, non-classical or variant cystic fibrosis, and pseudohypoaldosteronism
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2006-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
This is not an interventional study | This is not an interventional study
  Not applicable. This is not an interventional study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Knowles, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (9):
- United States (7):
  - Stanford University, Palo Alto, California
  - National Jewish Health, Denver, Colorado
  - The Children's Hospital, Denver, Colorado
  - Laboratory of Clinical Infectious Diseases, NIAID, Bethesda, Maryland
  - Washington University, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital and Regional Medical Center, Seattle, Washington
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Background] Kennedy MP, Ostrowski LE. Primary ciliary dyskinesia and upper airway diseases. Curr Allergy Asthma Rep. 2006 Nov;6(6):513-7. doi: 10.1007/s11882-006-0030-7. PMID 17026878
- [Background] Ferkol T, Leigh M. Primary ciliary dyskinesia and newborn respiratory distress. Semin Perinatol. 2006 Dec;30(6):335-40. doi: 10.1053/j.semperi.2005.11.001. PMID 17142159
- [Background] Zariwala MA, Knowles MR, Omran H. Genetic defects in ciliary structure and function. Annu Rev Physiol. 2007;69:423-50. doi: 10.1146/annurev.physiol.69.040705.141301. PMID 17059358
- [Background] Zariwala MA, Leigh MW, Ceppa F, Kennedy MP, Noone PG, Carson JL, Hazucha MJ, Lori A, Horvath J, Olbrich H, Loges NT, Bridoux AM, Pennarun G, Duriez B, Escudier E, Mitchison HM, Chodhari R, Chung EM, Morgan LC, de Iongh RU, Rutland J, Pradal U, Omran H, Amselem S, Knowles MR. Mutations of DNAI1 in primary ciliary dyskinesia: evidence of founder effect in a common mutation. Am J Respir Crit Care Med. 2006 Oct 15;174(8):858-66. doi: 10.1164/rccm.200603-370OC. Epub 2006 Jul 20. PMID 16858015
- [Background] Kennedy MP, Noone PG, Carson J, Molina PL, Ghio A, Zariwala MA, Minnix SL, Knowles MR. Calcium stone lithoptysis in primary ciliary dyskinesia. Respir Med. 2007 Jan;101(1):76-83. doi: 10.1016/j.rmed.2006.04.007. Epub 2006 Jun 6. PMID 16757159
- [Background] Hornef N, Olbrich H, Horvath J, Zariwala MA, Fliegauf M, Loges NT, Wildhaber J, Noone PG, Kennedy M, Antonarakis SE, Blouin JL, Bartoloni L, Nusslein T, Ahrens P, Griese M, Kuhl H, Sudbrak R, Knowles MR, Reinhardt R, Omran H. DNAH5 mutations are a common cause of primary ciliary dyskinesia with outer dynein arm defects. Am J Respir Crit Care Med. 2006 Jul 15;174(2):120-6. doi: 10.1164/rccm.200601-084OC. Epub 2006 Apr 20. PMID 16627867
- [Background] Horvath J, Fliegauf M, Olbrich H, Kispert A, King SM, Mitchison H, Zariwala MA, Knowles MR, Sudbrak R, Fekete G, Neesen J, Reinhardt R, Omran H. Identification and analysis of axonemal dynein light chain 1 in primary ciliary dyskinesia patients. Am J Respir Cell Mol Biol. 2005 Jul;33(1):41-7. doi: 10.1165/rcmb.2004-0335OC. Epub 2005 Apr 21. PMID 15845866
- [Background] Fliegauf M, Olbrich H, Horvath J, Wildhaber JH, Zariwala MA, Kennedy M, Knowles MR, Omran H. Mislocalization of DNAH5 and DNAH9 in respiratory cells from patients with primary ciliary dyskinesia. Am J Respir Crit Care Med. 2005 Jun 15;171(12):1343-9. doi: 10.1164/rccm.200411-1583OC. Epub 2005 Mar 4. PMID 15750039
- [Background] Zariwala MA, Despotes KA, Davis SD. Primary Ciliary Dyskinesia. 2007 Jan 24 [updated 2025 May 22]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1122/ PMID 20301301
- [Background] Kennedy MP, Noone PG, Leigh MW, Zariwala MA, Minnix SL, Knowles MR, Molina PL. High-resolution CT of patients with primary ciliary dyskinesia. AJR Am J Roentgenol. 2007 May;188(5):1232-8. doi: 10.2214/AJR.06.0965. PMID 17449765
- [Background] Morillas HN, Zariwala M, Knowles MR. Genetic causes of bronchiectasis: primary ciliary dyskinesia. Respiration. 2007;74(3):252-63. doi: 10.1159/000101783. PMID 17534128
- [Background] Kennedy MP, Omran H, Leigh MW, Dell S, Morgan L, Molina PL, Robinson BV, Minnix SL, Olbrich H, Severin T, Ahrens P, Lange L, Morillas HN, Noone PG, Zariwala MA, Knowles MR. Congenital heart disease and other heterotaxic defects in a large cohort of patients with primary ciliary dyskinesia. Circulation. 2007 Jun 5;115(22):2814-21. doi: 10.1161/CIRCULATIONAHA.106.649038. Epub 2007 May 21. PMID 17515466
- [Background] Loges NT, Olbrich H, Becker-Heck A, Haffner K, Heer A, Reinhard C, Schmidts M, Kispert A, Zariwala MA, Leigh MW, Knowles MR, Zentgraf H, Seithe H, Nurnberg G, Nurnberg P, Reinhardt R, Omran H. Deletions and point mutations of LRRC50 cause primary ciliary dyskinesia due to dynein arm defects. Am J Hum Genet. 2009 Dec;85(6):883-9. doi: 10.1016/j.ajhg.2009.10.018. PMID 19944400
- [Background] Leigh MW, Pittman JE, Carson JL, Ferkol TW, Dell SD, Davis SD, Knowles MR, Zariwala MA. Clinical and genetic aspects of primary ciliary dyskinesia/Kartagener syndrome. Genet Med. 2009 Jul;11(7):473-87. doi: 10.1097/GIM.0b013e3181a53562. PMID 19606528
- [Result] Zariwala MA, Omran H, Ferkol TW. The emerging genetics of primary ciliary dyskinesia. Proc Am Thorac Soc. 2011 Sep;8(5):430-3. doi: 10.1513/pats.201103-023SD. PMID 21926394
- [Result] Leigh MW, O'Callaghan C, Knowles MR. The challenges of diagnosing primary ciliary dyskinesia. Proc Am Thorac Soc. 2011 Sep;8(5):434-7. doi: 10.1513/pats.201103-028SD. PMID 21926395
- [Result] Sagel SD, Davis SD, Campisi P, Dell SD. Update of respiratory tract disease in children with primary ciliary dyskinesia. Proc Am Thorac Soc. 2011 Sep;8(5):438-43. doi: 10.1513/pats.201103-024SD. PMID 21926396
- [Result] Davis SD, Knowles M, Leigh M. Introduction: primary ciliary dyskinesia and overlapping syndromes. Proc Am Thorac Soc. 2011 Sep;8(5):421-2. doi: 10.1513/pats.201103-026SD. No abstract available. PMID 21926392
- [Result] Mateos-Corral D, Coombs R, Grasemann H, Ratjen F, Dell SD. Diagnostic value of nasal nitric oxide measured with non-velum closure techniques for children with primary ciliary dyskinesia. J Pediatr. 2011 Sep;159(3):420-4. doi: 10.1016/j.jpeds.2011.03.007. Epub 2011 Apr 22. PMID 21514598
- [Result] Knowles MR, Leigh MW, Carson JL, Davis SD, Dell SD, Ferkol TW, Olivier KN, Sagel SD, Rosenfeld M, Burns KA, Minnix SL, Armstrong MC, Lori A, Hazucha MJ, Loges NT, Olbrich H, Becker-Heck A, Schmidts M, Werner C, Omran H, Zariwala MA; Genetic Disorders of Mucociliary Clearance Consortium. Mutations of DNAH11 in patients with primary ciliary dyskinesia with normal ciliary ultrastructure. Thorax. 2012 May;67(5):433-41. doi: 10.1136/thoraxjnl-2011-200301. Epub 2011 Dec 18. PMID 22184204
- [Result] Stillwell PC, Wartchow EP, Sagel SD. Primary Ciliary Dyskinesia in Children: A Review for Pediatricians, Allergists, and Pediatric Pulmonologists. Pediatr Allergy Immunol Pulmonol. 2011 Dec;24(4):191-196. doi: 10.1089/ped.2011.0099. PMID 22276227
- [Result] Knowles MR, Leigh MW, Zariwala MA. Cutting edge genetic studies in primary ciliary dyskinesia. Thorax. 2012 May;67(5):464; author reply 464. doi: 10.1136/thoraxjnl-2012-201609. Epub 2012 Feb 10. No abstract available. PMID 22328589
- [Result] Ferkol TW, Leigh MW. Ciliopathies: the central role of cilia in a spectrum of pediatric disorders. J Pediatr. 2012 Mar;160(3):366-71. doi: 10.1016/j.jpeds.2011.11.024. Epub 2011 Dec 16. No abstract available. PMID 22177992
- [Result] Nakhleh N, Francis R, Giese RA, Tian X, Li Y, Zariwala MA, Yagi H, Khalifa O, Kureshi S, Chatterjee B, Sabol SL, Swisher M, Connelly PS, Daniels MP, Srinivasan A, Kuehl K, Kravitz N, Burns K, Sami I, Omran H, Barmada M, Olivier K, Chawla KK, Leigh M, Jonas R, Knowles M, Leatherbury L, Lo CW. High prevalence of respiratory ciliary dysfunction in congenital heart disease patients with heterotaxy. Circulation. 2012 May 8;125(18):2232-42. doi: 10.1161/CIRCULATIONAHA.111.079780. Epub 2012 Apr 12. PMID 22499950
- [Result] Horani A, Druley TE, Zariwala MA, Patel AC, Levinson BT, Van Arendonk LG, Thornton KC, Giacalone JC, Albee AJ, Wilson KS, Turner EH, Nickerson DA, Shendure J, Bayly PV, Leigh MW, Knowles MR, Brody SL, Dutcher SK, Ferkol TW. Whole-exome capture and sequencing identifies HEATR2 mutation as a cause of primary ciliary dyskinesia. Am J Hum Genet. 2012 Oct 5;91(4):685-93. doi: 10.1016/j.ajhg.2012.08.022. PMID 23040496
- [Result] Ferkol TW, Puffenberger EG, Lie H, Helms C, Strauss KA, Bowcock A, Carson JL, Hazucha M, Morton DH, Patel AC, Leigh MW, Knowles MR, Zariwala MA. Primary ciliary dyskinesia-causing mutations in Amish and Mennonite communities. J Pediatr. 2013 Aug;163(2):383-7. doi: 10.1016/j.jpeds.2013.01.061. Epub 2013 Mar 7. PMID 23477994
- [Derived] Kaspy KR, Dell SD, Davis SD, Ferkol TW, Rosenfeld M, Sagel SD, Milla C, Olivier KN, Barber AT, Wee W, Lin FC, Li L, Rampakakis E, Zariwala MA, Knowles MR, Leigh MW, Shapiro AJ. Situs Ambiguus Is Associated With Adverse Clinical Outcomes in Children With Primary Ciliary Dyskinesia. Chest. 2024 May;165(5):1070-1081. doi: 10.1016/j.chest.2023.12.005. Epub 2023 Dec 9. PMID 38072392
- [Derived] Leigh MW, Ferkol TW, Davis SD, Lee HS, Rosenfeld M, Dell SD, Sagel SD, Milla C, Olivier KN, Sullivan KM, Zariwala MA, Pittman JE, Shapiro AJ, Carson JL, Krischer J, Hazucha MJ, Knowles MR. Clinical Features and Associated Likelihood of Primary Ciliary Dyskinesia in Children and Adolescents. Ann Am Thorac Soc. 2016 Aug;13(8):1305-13. doi: 10.1513/AnnalsATS.201511-748OC. PMID 27070726
- [Derived] Shapiro AJ, Davis SD, Ferkol T, Dell SD, Rosenfeld M, Olivier KN, Sagel SD, Milla C, Zariwala MA, Wolf W, Carson JL, Hazucha MJ, Burns K, Robinson B, Knowles MR, Leigh MW; Genetic Disorders of Mucociliary Clearance Consortium. Laterality defects other than situs inversus totalis in primary ciliary dyskinesia: insights into situs ambiguus and heterotaxy. Chest. 2014 Nov;146(5):1176-1186. doi: 10.1378/chest.13-1704. PMID 24577564